CLINICAL TRIAL: NCT06539338
Title: A Two-Part Open Label Phase 1 Multicentre Study Evaluating the Safety of INT2104 Infusion in Female and Male Participants Aged 18 Years of Age and Older With Refractory/Relapsing B-Cell Malignancies
Brief Title: A Study to Investigate Safety of INT2104 Infusions in Participants Aged 18 Years of Age and Older Who Have B-cell Cancers That Came Back After Previous Treatment
Acronym: INVISE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INT2104-101; 2023-509132-26-00 (EU CTIS Number); U1111-1303-9462 (Other: WHO)
Record Dates: First submitted 2024-06-19; First posted 2024-08-06 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Lymphomas Non-Hodgkin's B-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma
Keywords: Gene Therapy
MeSH Terms: conditions — Lymphoma, B-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- INT2104 Dose Level 1 (Experimental): Single IV administration of INT2104
  Interventions: Genetic: INT2104
- INT2104 Dose Level 2 (Experimental): Single IV administration of INT2104
  Interventions: Genetic: INT2104
- INT2104 Dose Level 3 (Experimental): Single IV administration of INT2104
  Interventions: Genetic: INT2104
- INT2104 Dose Level 4 (Experimental): Single IV administration of INT2104
  Interventions: Genetic: INT2104
- INT2104 Recommended Dose (Experimental): Single IV administration of INT2104
  Interventions: Genetic: INT2104

INTERVENTIONS:
Genetic: INT2104 — INT2104 is a lentiviral vector delivering a transgene for a chimeric antigen receptor specific for CD20 (CAR20)

SUMMARY:
The purpose of this first-in-human study is to evaluate the safety and tolerability of INT2104 when administered to humans in a broad population of participants with refractory/relapsing B-cell malignancies. Preliminary efficacy information may also be obtained.

INT2104 is a gene therapy delivering a transgene for a chimeric antigen receptor (CAR) specific for CD20 (CAR20). The lentiviral vector is designed to generate CAR T and CAR Natural Killer (NK) cells inside the body following intravenous (IV) administration.

Study details include the following:

* The study duration will be 5 years
* The treatment duration will be a one-time intravenous (IV) infusion of INT2104

DETAILED DESCRIPTION:
This is a non-randomized, open label, multi-site, Phase 1 First in Human (FIH) study split into two parts. The first part (Part A) is a dose escalation and the second part (Part B) will be to confirm the dose.

The aim of the study is to collect data to assess whether the study product, INT2104, is safe and tolerable, to understand how well INT2104 works in the human body and to select the dose to take into a Phase 2 study.

All participants will receive one intravenous (IV) infusion of INT2104.

Each participant in the study will follow the same study treatment schedule and will proceed through the following study periods:

* Screening Period: participant will be assessed for eligibility
* Study Day 1: participants who meet all eligibility criteria will receive INT2104 by a one-time infusion
* Post-treatment Assessment Period: participants will be followed regularly with clinic visits after they receive INT2104

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with relapsed/refractory (R/R) B-NHL (Burkitt's lymphoma are eligible for Part B only) confirmed by histology or flow cytometry Note: Bone Marrow involvement is allowed
* B-NHL must have CD20 antigen positive tumour confirmed from a tumour biopsy taken at screening
* Measurable disease at the time of enrolment
* Progression after at least 2 lines of systemic therapy
* Has not received more than one prior marketed CAR-T cell therapy (including tandem or bispecific CAR-T) or other genetically modified T-cell therapy.
* Sex and Contraceptive/Barrier Requirements consistent with local regulations for clinical trials Females: must have negative serum pregnancy test at screening and on Day -1 prior to INT2104 infusion Both sexes: must agree to use highly effective methods, including a barrier method after INT2104 infusion
* Haematological criteria:

  * Absolute lymphocyte count (ALC) ≥300/µL
  * Platelet count ≥50,000/mL
  * Absolute neutrophil count (ANC) ≥500/µL
* Eastern Cooperative Oncology Group (ECOG) score of 0 or 1
* Adequate renal, cardiac, hepatic, and lung function

Key Inclusion Part B only

* Diagnosed with relapsed/refractory B-ALL, and with exceptions as detailed in exclusion criteria. Participants with Philadelphia chromosome positive (Ph+) B-ALL disease are eligible.
* B-ALL participants must have CD20 antigen positive leukaemia
* Measurable disease at the time of enrolment
* Participants with Burkitt's lymphoma are eligible for Part B only

Exclusion Criteria:

* Central Nervous System (CNS)-only B-cell malignancy, or B-cell malignancy with R/R secondary CNS involvement.
* Diagnosis or history of chronic lymphocytic leukaemia (CLL) (including large cell [Richter] transformation of CLL) or small lymphocytic lymphoma (SLL)
* Diagnosis or history of cutaneous lymphoma
* History of another primary malignancy that has not been in remission for at least 3 years before signing informed consent (except for: non-melanoma skin cancer, low grade prostate cancer or carcinoma in situ (e.g., cervix, bladder, breast))
* Acute or chronic graft-versus-host disease
* Participant has received donor lymphocyte infusion within 6 weeks prior to INT2104 infusion
* History of autoimmune disease requiring systemic immunosuppression/ systemic disease modifying agents within 2 years before enrolment
* History or presence of CNS disorder
* History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months before signing informed consent
* Participants has active syphilis, cytomegalovirus (CMV), acute or chronic active hepatitis B, or untreated hepatitis C.
* Participant is Human immunodeficiency virus (HIV) positive.
* Any medical condition likely to interfere with assessment of safety or efficacy of the study treatment
* A vaccine within 4 weeks prior to INT2104 infusion
* Intolerance or severe hypersensitivity reaction to any excipients of the INT2104 product.
* An active fungal, bacterial, viral, or other infection that is uncontrolled or requires antimicrobials at the time of INT2104 infusion.
* Participant is pregnant or nursing.
* In the investigator's judgment, the participant is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events | Up to 5 years
  Number of Participants With Adverse Events as Assessed by CTCAE v5.0
Number of Participants With Abnormal Clinical Laboratory Values and Physical Examination Results | Baseline, up to Day 29
  Number of Participants With abnormal clinical laboratory values as Assessed by CTCAE v5.0
Number of Participants Experiencing Cytokine Release Syndrome (CRS) | Baseline, up to Day 29
  Number of participants experiencing Cytokine Release Syndrome (CRS)
Number of Participants Experiencing Immune Effector Cell Neurotoxicity (ICANS) | 28 Days
  Number of participants experiencing Immune Effector Cell Neurotoxicity (ICANS)
Number of Participants Experiencing dose-limiting toxicities (DLTs) | 28 Days
  Number of participants experiencing dose-limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Levels of Vector Ribonucleic Acid (RNA) Genomes in Blood Over Time | Baseline, up to Day 29
Levels of Transgene Deoxyribonucleic Acid (DNA) Copies in Blood Over Time | Baseline, up to Day 29
Levels of CD20-targeting Chimeric Antigen Receptor (CAR20) Positive T Cells in Blood Over Time | Baseline, up to Day 29
Levels of Natural Killer (NK) Cells in Blood Over Time | Baseline, up to Day 29
Number of Participants with CAR20-positive Cells in Accessible Tumour Tissue Over Time | Baseline, up to Day 29
Change in the Levels of Lymphocyte Subsets Including B-cell Counts Over Time | Baseline, up to Day 29
Objective Response Rate (ORR) as Determined by Investigator Assessment | Day 90
Objective Response Rate (ORR) as Determined by Investigator Assessment | Year 1
Objective Response Rate (ORR) as Determined by Investigator Assessment | Year 2
Objective Response Rate (ORR) as Determined by Investigator Assessment | Year 5
Complete Response (CR) Rate as Determined by Investigator Assessment | Day 90
Complete Response (CR) Rate as Determined by Investigator Assessment | Year 1
Complete Response (CR) Rate as Determined by Investigator Assessment | Year 2
Complete Response (CR) Rate as Determined by Investigator Assessment | Year 5
Duration of response (DOR) as Determined by Investigator Assessment | Up to 5 years
Progression Free Survival (PFS) as Determined by Investigator Assessment | Up to 5 years
Overall Survival (OS) as Determined by Investigator Assessment | Up to 5 years
Number of Participants with Cytokine Release Syndrome (CRS) | Up to 5 years
Number of Participants with Immune Effector Cell-associated Neurotoxicity Syndrome (ICANS) | Up to 5 years
Duration of Cytokine Release Syndrome (CRS) | Up to 5 years
Duration of ICANS | Up to 5 years
Number of Participants with Vector-derived Replication Competent Lentivirus (RCL) Through Year 5 | Up to 5 years
Assessment of Humoral Immunity: Number of Participants with Anti-CAR and Anti-vector Antibodies Over Time | Up to 5 years
Assessment of Cellular Immunity: Number of Participants with Changes in T-cell Enzyme-Linked Immunospot Assay (ELISPOT) and Cytokine Profiles Over Time | Up to 5 years
Assessment of Vector Shedding: Number of Participants with Vector Shedding in Saliva, Faeces, and Urine Over Time | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (3):
- Australia (2):
  - Westmead Hospital, Westmead, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Hospital MD Anderson, Madrid, Spain

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06539338